CLINICAL TRIAL: NCT06637943
Title: Comparison of Time Taken for Diagnosing Intraoperative Coagulopathies: Point-of-care Viscoelastic Tests vs Standard Central Laboratory Tests
Brief Title: Comparison of the Diagnosis Time of VET and SCL in Patients With Intraoperative Coagulopathy
Status: Not yet recruiting | Type: Observational
Sponsor: Konkuk University Medical Center (Other)
Collaborators: Korea Health Industry Development Institute (Other Government); Asan Medical Center (Other); Samsung Medical Center (Other); Soon Chun Hyang University (Other)
Responsible Party: Principal Investigator, Tae-Yop Kim, MD PhD, Professor of Anesthesiology, Konkuk University Medical Center
Other Study IDs: HI22C1952-1-2-2
Record Dates: First submitted 2024-10-07; First posted 2024-10-15 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Arthritis of Knee; Arthritis of Hip; Spine; Prostate Cancer; Hepatic Cancer; Valvular Disorder; Ischemic Heart Disease; Aortic Diseases
Keywords: viscoelastic test; standard central laboratory test; coagulation
MeSH Terms: conditions — Prostatic Neoplasms; Liver Neoplasms; Myocardial Ischemia; Aortic Diseases; Thrombosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SCL tests: standard central laboratory (SCL) tests
  Interventions: Diagnostic Test: SCL tests
- POC viscoleastic tests: point-of-care (POC) viscoelastic tests
  Interventions: Diagnostic Test: POC viscoelastic tests

INTERVENTIONS:
Diagnostic Test: SCL tests — applying PT-INR, serum-fibrinogen (Claus Method), serum-platelet count
  Groups: SCL tests
Diagnostic Test: POC viscoelastic tests — applying ROTEM or TEG
  Groups: POC viscoleastic tests

SUMMARY:
The present study is a prospective, multi-center observational trial comparing the times taken to diagnose coagulopathies using point-of-care (POC) viscoelastic tests or standard central laboratory tests (SCL tests) in patients with intraoperative bleeding.

DETAILED DESCRIPTION:
The present study is a prospective multi-center observational trial comparing the time for diagnosing coagulopathies using POC viscoelastic tests, such as rotational thromboelastometry (ROTEM) and thromboelastography (TEG) and standard central laboratory tests (SCL test, such as PT-INR, aPTT, s-fibrinogen level, platelet count) in intraoperative bleeding patients.

The study will be performed during surgeries that are expected to entail a moderate to severe amount of bleeding and warrant the use of either POC viscoelastic tests, SCL tests, or both to determine the possible association of coagulopathy.

The tests will be conducted when an intraoperative condition requires identifying possible associations of coagulopathies during and after surgical bleeding. The test results will prompt appropriate coagulation management.

The primary objective is to compare the diagnosis time for intraoperative coagulopathy using the POC viscoelastic test or SCL test. The time will be defined as the time elapsed from the time obtaining a blood sample for the POC viscoelastic test or SCL test to the time acknowledging the test results.

Researchers hypothesized that using POC viscoelastic tests would shorten the time for diagnosis compared to SCL tests.

ELIGIBILITY:
Inclusion Criteria:

* patients who will undergo elective surgery with a high risk of moderate to severe amount of intraoperative bleeding or coagulopathy (e.g., cardiac surgery, joint replacement, spine surgery, hepatectomy, radical prostatectomy)
* patients who provide written informed consent
* patients who may warrant the intraoperative use of POC viscoelastic test or SCL test

Exclusion Criteria:

* pregnancy
* withdrawal of consent
* termination of surgery without performing either POC viscoelastic test or SCL tests
* when the study conductor deems it inappropriate to proceed with the protocol with the patient

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: conditions/ diseases
  * Arthritis of knee
  * Arthritis of hip
  * Spine
  * Prostate cancer
  * Hepatic cancer
  * Valvular dysfunction
  * Ischemic heart disease
  * Aortic disease
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Time for establishing a diagnosis using viscoelastic test and SCL test, minute | From the start and to the end of surgery, an average of 6 hours
  Lapsed time (minute) from obtaining a blood sample to identifying association or absence of coagulation dysfunction

SECONDARY OUTCOMES:
Test results from viscoelastic test and SCL test | From the start and to the end of surgery, an average of 6 hours
  ROTEM (CT-EXTEM, A5-EXTEM, A10-EXTEM, A15-EXTEM, MCF-EXTEM, A5-FIBTEM, A10-FIBTEM, MCF-FIBTEM), TEG (CK R-time, CK alpha angle CRT MA, CFF MA), SCL (hemoglobin, PT-INR, aPTT, platelet count, serum-fibrinogen level) The test results for deciding to give PRBCs: hemoglobin value (g/dl) in both groups The test results for deciding to give FFPs: CT-EXTEM (mm) in the study group vs PT-INR in the control group The test results for deciding to give cryoprecipitates: A5-FIBTEM or MCF-FIBTEM (mm) in the study group vs serum fibrinogen level (mg/dl) in the control group The test results for deciding to give platelets: A5-PLETEM (A5-EXTEM, A5-FIBTEM. mm) or MCF-PLTEM (MCF-EXTEM, MCF-FIBTEM, mm) in the study group vs serum-fibrinogen level (mg/dl) in the control group
The difference in the percentages of patients that lead to the diagnosis of coagulopathies for viscoelastic test and SCL tests | From the start and to the end of surgery, an average of 6 hours
  The difference in the percentages of patients that lead to the diagnosis of coagulopathies for viscoelastic test and SCL tests, respectively, when both tests were performed simultaneously
Time for initiating a treatment, munute | From the start and to the end of surgery, an average of 6 hours
  Defined as lapsed time from acknowledging the result of the test and ordering blood products if indicated (minute)
Time taken to complete the delivery of the blood products to the operation room, minute | From the start and to the end of surgery, an average of 6 hours
  Time taken to complete the delivery of the blood products to the operation room, minute
Amount of blood products transfused if indicated specific to each test, unit | From the start and to the end of surgery, an average of 6 hours
  Amount of blood products transfused if indicated specific to each test packed red blood cells (PRBCs), fresh frozen plasma (FFP), cryoprecipitate, platelet (unit)
comparisons of diagnosis time between POC-viscoelastic test and SCL test | From the start and to the end of surgery, an average of 6 hours
  Lapsed time (minutes) from obtaining a blood sample to identifying the association or absence of coagulation dysfunction in the POC viscoelastic tests and SCL tests

CONTACTS AND LOCATIONS:
Overall Officials: Tae-Yop Kim, MD, PhD, Principal Investigator — Konkuk University Medical Center
Locations (4):
- South Korea (4):
  - Asan Medical Center, Seoul, Seoul
  - Konkuk Univeristy Medical Center, Seoul, Seoul
  - Samsung Medical Center, Seoul
  - Sooncheonhyang University, Seoul

IPD SHARING:
Plan to Share IPD: Undecided